CLINICAL TRIAL: NCT01324531
Title: Arthroscopic Bankart Repair With and Without Arthroscopic Infraspinatus Remplissage in Anterior Shoulder Instability With a Hill-Sachs Defect: A Randomized Controlled Trial
Brief Title: Arthroscopic Bankart Repair With and Without Remplissage in Anterior Shoulder Instability
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: University of Ottawa (Other); Western University, Canada (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Department Head, Orthopaedic Surgery, Panam Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REMP 01
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Other Instability, Shoulder; Hill-Sachs Lesion
Keywords: Bankart repair; remplissage; Hill-Sachs defect; shoulder instability; anterior shoulder instability
MeSH Terms: conditions — Bankart Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bankart repair (Active Comparator)
  Interventions: Procedure: Bankart repair
- Bankart repair and remplissage (Active Comparator)
  Interventions: Procedure: Bankart repair and remplissage

INTERVENTIONS:
Procedure: Bankart repair and remplissage — Bankart repair may be completed before or after remplissage. While maintaining camera in anterior-superior portal drill guide and anchor cannula is placed through the posterior portal into remplissage site. Anchor cannula with obturator is passed through infraspinatus tendon and posterior capsule via pre-existing portal, and first anchor is placed in inferior aspect of Hill-Sachs lesion.Once anchor is inserted, penetrating grasper is passed through tendon and posterior capsule, 1 cm inferior to the initial portal entry site, to grasp and pull 1 suture limb.Second anchor is placed in superior aspect of Hill-Sachs lesion and grasper penetrator is used in same fashion to pass 1 suture limb 1 cm superior to initial portal entry site. The inferior suture is tied first with knots remaining extraarticular in the subdeltoid space. The superior suture is tied to complete remplissage.
  Arms: Bankart repair and remplissage
Procedure: Bankart repair — Bankart repair based on surgeon's preference
  Arms: Bankart repair

SUMMARY:
The purpose of this prospective, randomized, controlled trial is to compare subjective patient-reported outcomes and objective clinical results between arthroscopic Bankart repair with and without arthroscopic infraspinatus remplissage in patients with anterior shoulder instability with a Hill-Sachs Defect.

DETAILED DESCRIPTION:
Significant osseous defects of the glenohumeral joint can often lead to failure of arthroscopic shoulder stabilization procedures. The best treatment in the setting of shoulder instability with significant glenoid and/or humeral defects remains controversial. Several open procedures have been suggested, but arthroscopic methods have started to garner some attention in the literature. In patients with an engaging Hill-Sachs lesion without significant glenoid bone loss, arthroscopic remplissage consisting of arthroscopic posterior capsulodesis and infraspinatus tenodesis to fill the Hill-Sachs lesion has been proposed as a novel treatment method.

The authors believe it is scientifically necessary to investigate the role of addition of arthroscopic infraspinatus remplissage to the conventional arthroscopic Bankart repair. As more surgeons are trained in the technique, it will be performed more frequently. Increased patient awareness continues to lead to increasing demand for minimally invasive approaches. Arthroscopic remplissage brings with it an increase in operative time, with a theorized risk of reduction in dislocation risk. For these reasons, the authors believe that it is scientifically and fiscally necessary to determine the difference in outcome between arthroscopic Bankart repair with and without arthroscopic infraspinatus remplissage for patients with anterior shoulder instability and a Hill-Sachs defect in the framework of a prospective, randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* 14 years or older
* must have anterior shoulder instability and Hill-Sachs defect
* must have anterior instability with any engaging Hill Sachs Lesion on CT scan, MRI or ultrasound and no more than 15% glenoid bone loss

Exclusion Criteria:

* Glenoid defect >15% of AP diameter of glenoid
* significant shoulder comorbidities (i.e, OA, previous surgery other than previous instability)
* active joint or systemic infection
* significant muscle paralysis
* rotator cuff or Charcot's arthropathy
* significant medical comorbidity that may alter effectiveness of surgical intervention
* major medical illness
* unable to speak French or English
* psychiatric illness that precludes informed consent
* unwilling to be followed for 2 years

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2019-06 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability (WOSI) score | 24 months post-surgery
  WOSI score questionnaire is a tool designed for self-assessment of shoulder function for patients with instability problems. Difference between study arm outcomes will be assessed using pre-op WOSI score as a covariate

SECONDARY OUTCOMES:
Simple Shoulder Test | 24 months post-surgery
  Simple Shoulder Test (SST) is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment. Differences between study arm outcomes will be assessed using pre-op SST scores as a covariate
American Shoulder and Elbow Society assessment (ASES) | 24 months post-surgery
  The ASES assessment (patient report section) is a region-specific questionnaire designed for self-assessment of aspects of pain and function. Difference between study arm outcomes will be assessed using pre-op ASES score as a covariate
Ultrasound imaging | 24 months post-surgery
  Ultrasound imaging will be conducted 24 months post-surgery and compared to pre-operative findings on CT-Scan, ultrasound and intraoperatively to establish extent of healing.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Pan Am Clinic, Winnipeg, Manitoba
  - University of Ottawa/Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Background] Burkhart SS, De Beer JF. Traumatic glenohumeral bone defects and their relationship to failure of arthroscopic Bankart repairs: significance of the inverted-pear glenoid and the humeral engaging Hill-Sachs lesion. Arthroscopy. 2000 Oct;16(7):677-94. doi: 10.1053/jars.2000.17715. PMID 11027751
- [Background] Burkhart SS, Danaceau SM. Articular arc length mismatch as a cause of failed bankart repair. Arthroscopy. 2000 Oct;16(7):740-4. doi: 10.1053/jars.2000.7794. PMID 11027759
- [Background] Kropf EJ, Tjoumakaris FP, Sekiya JK. Arthroscopic shoulder stabilization: is there ever a need to open? Arthroscopy. 2007 Jul;23(7):779-84. doi: 10.1016/j.arthro.2007.03.004. PMID 17637415
- [Derived] Woodmass JM, McRae S, Lapner P, Kamikovski I, Jong B, Old J, Marsh J, Dubberley J, Stranges G, Sasyniuk TM, MacDonald PB. Arthroscopic Bankart Repair With Remplissage in Anterior Shoulder Instability Results in Fewer Redislocations Than Bankart Repair Alone at Medium-term Follow-up of a Randomized Controlled Trial. Am J Sports Med. 2024 Jul;52(8):2055-2062. doi: 10.1177/03635465241254063. Epub 2024 Jun 14. PMID 38874505